CLINICAL TRIAL: NCT03020355
Title: Comparison of Blood Loss in Using vs Not Using Placental Cord Drainage After Spontaneous Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, Medical Doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 167
Record Dates: First submitted 2016-12-22; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Placental Blood Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placental Blood Drainage (Experimental): Immediately after vaginal delivery, after clamping and cutting the cord-the cord will unclamped and the blood will drained until the flow ceased.
  Interventions: Procedure: Placental Blood Drainage
- not Placental Blood Drainage (Active Comparator): In the control group, the clamped cord will not released.
  Interventions: Procedure: not Placental Blood Drainage

INTERVENTIONS:
Procedure: Placental Blood Drainage — Immediately after vaginal delivery, after clamping and cutting the cord-the cord will unclamped and the blood will drained until the flow ceased.
  Arms: Placental Blood Drainage
Procedure: not Placental Blood Drainage — In the control group, the clamped cord will not released.
  Arms: not Placental Blood Drainage

SUMMARY:
Comparison of effectiveness of placental blood drainage after spontaneous vaginal delivery in decreasing the duration, blood loss,and complications of the third stage, against no drainage of placental blood.

DETAILED DESCRIPTION:
The patients will prospectively randomized equally into two groups (100 each in the study and control groups).

Group-A (Study group)-Placental blood was drained.

Group-B (Control group)-Placental blood was not drained.

In all the patients detailed medical and obstetric history will taken. In each patient, the pre-delivery pulse rate, blood pressure, and Hb gm% will noted. Immediately after vaginal delivery, after clamping and cutting the cord-the cord will unclamped and the blood will drained until the flow ceased. In the control group, the clamped cord will not released. Blood lost in the third stage of labour will measured by collecting the blood measuring bag.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Vertex presentation
* Gestational age of 37 weeks (or) more
* No major medical (or) obstetric complications
* Spontaneous vaginal delivery

Exclusion Criteria:

* Hb\7 gm/dl
* History of APH
* Instrumental delivery
* Multiple pregnancy
* Malpresentations
* Large baby (more than 3.5 kg)
* Polyhydramnios
* Known coagulations disorders
* Previous surgeries on the uterus

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Blood lost | through delivery completion, an average of 30 minutes

SECONDARY OUTCOMES:
The duration of the third stage | through the duration of the third stage, an average 45 minutes
  The duration of the third stage will calculated using a stop watch.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Roy P, Sujatha MS, Bhandiwad A, Biswas B, Chatterjee A. Placental Blood Drainage as a Part of Active Management of Third Stage of Labour After Spontaneous Vaginal Delivery. J Obstet Gynaecol India. 2016 Oct;66(Suppl 1):242-5. doi: 10.1007/s13224-016-0857-3. Epub 2016 Mar 12. PMID 27651611
- [Result] Soltani H, Poulose TA, Hutchon DR. Placental cord drainage after vaginal delivery as part of the management of the third stage of labour. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD004665. doi: 10.1002/14651858.CD004665.pub3. PMID 21901693